CLINICAL TRIAL: NCT03102827
Title: High-Flow-Therapy for the Treatment of Cheyne-Stokes-Respiration in Chronic Heart Failure
Acronym: FLOAT-CS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unavailability of PI and Deputy
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Thomas Bitter, Senior physician, Heart and Diabetes Center North-Rhine Westfalia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HDZNRW-KA_006-TB
Record Dates: First submitted 2017-03-21; First posted 2017-04-06 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure | interventions — Oxygen; Particulate Matter

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen - ambient air (Active Comparator): high-flow oxygen therapy administered during first night, ambient air without high-flow therapy (placebo) administered during second night
  Interventions: Drug: Oxygen
- Ambient air - oxygen (Placebo Comparator): Ambient air without high-flow therapy (placebo) administered during first night , high-flow oxygen therapy administered during second night
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxygen — Patients will receive oxygen with humidified air, fully saturated at 37° C at a flow rate of 20- 50 L/min. The ratio of oxygen and ambient air (FiO2) will be increased stepwise depending on patient's oxygen saturation.
  Other Names: CONOXIA® GO2X
  Arms: Oxygen - ambient air
Other: Placebo — Ambient air without high-flow therapy administered during first night
  Other Names: Ambient air
  Arms: Ambient air - oxygen

SUMMARY:
To demonstrate the effectiveness and safety of nocturnal ventilation with oxygen (HFT - high-flow-therapy) for the treatment of CSA in patients with HFrEF compared to placebo (patient will breathe ambient air via nasal cannula that is not connected to the high-flow-device).

DETAILED DESCRIPTION:
In chronic heart failure (CHF) patients sleep disordered breathing mainly comprises two different entities: obstructive sleep apnea (OSA) and central sleep apnea with Cheyne-Stokes respiration (CSA). Being a rare disease in the general population, CSA is found with a prevalence of up to 40% in CHF patients.1 This rise in prevalence is instigated by pathophysiological overlapses. CSA is precipitated by hyperventilation and a highly sensitive hypocapnea-induced apneic threshold, whereby apnea is then initiated by small transient reductions in partial pressure of carbon dioxide (pCO2). Underlying mechanisms are not fully understood, yet. Despite neurohumoral derangement such as altered chemoreflex cascades (enhanced "loop gain" and "controller gain") and circulatory delay, pulmonary congestion is thought to play a role in the evolution of CSA. Caused by reduced cardiac output and/or impaired left ventricular filling pattern, a rise in pulmonary capillary wedge pressure (PCWP) with resulting interstitial pulmonary edema is closely correlated to the occurrence of CSA. Furthermore, acute increase in pulmonary congestion by overnight rostral fluid displacement to the lungs was found to lower sleep pCO2 and predisposed to CSA. Furthermore, decreased blood oxygen tension stimulates the discharge of peripheral chemoreceptors and gives rise to hyperventilation pattern of CSA. Conversely, hyperventilation increases the propensity for central apneas by reducing the CO2-reserve. Underlining the importance of hypoxemic chemoreceptor stimulation in the development of CSA, previous studies exemplified this as a pathophysiological key element in patient with pulmonary artery hypertension, where hypocapnia, periodic breathing and CSA is highly prevalent despite normal capillary wedge pressure values. Also in heart failure patients this seems to be important: several interventional studies showed an at least partial suppression of CSR using oxygen therapy.

High flow therapy is a technique that provides a range of flows of heated, humidified air to patients requiring respiratory support, delivered through nasal cannula range The high flow ventilation therapy with an air/oxygen mixture at a rate of 20-50 L/min via a nasal cannula is able to provide adequate oxygen flow rates to completely avoid hypoxemias. An increase in oxygen saturation is associated with a reduced chemosensitivity of the glomus caroticum. This may further help to improve Cheyne-Stokes respiration severity. Previous studies could reach a reduction of 50% of the AHI with the use of 2 L/min of oxygen.

At the same time the high flow ventilation therapy can attenuate inspiratory resistance by potentially delivering positive distending pressure for lung recruitment without providing excessive intrathoracic pressure (only 3-6 cm H2O, according to manufacturer).

But on the other hand the hyperoxemic state was also found to have some unfavorable consequences such as an increase in infarct size after myocardial infarction and should therefore be avoided.

The FLOAT-CS study is a proof-of-concept study that investigates nocturnal high flow ventilation therapy with oxygen (oxygen-HFT) as a novel therapeutic approach for HFrEF patients with CSA by attenuation of the hypoxemic burden.

The high flow ventilation therapy via a nasal cannula with 20-50 L/min of a mixture of ambient air and oxygen is titrated to achieve a target oxygen flow that leads to normoxemia defined as a transcutaneous oxygen saturation (SpO2) between 91% and 98%. This is expected to completely avoid hypoxemias without providing excessive intrathoracic pressure. For the greatest possible comfort of the patients a humidifier is used and the mixture of air and oxygen is warmed up to 37°C.

In addition, the FLOAT-CS study investigates the hemodynamic effects of oxygen-HFT versus placebo.

Thus the patients participating in the study are randomized in a 1:1 manner to therapy with oxygen-HFT either during their first or their second study night, respectively. During the other night they are treated with placebo.

Since the main focus of this investigation is treatment of CSA patients will undergo fully-attended, in-hospital polysomnography to assess parameters related to sleep and cardiorespiratory events during sleep All subjects receive an arterial access of the Arteria radialis that remains throughout their study participation. This allows for a continuous invasive hemodynamic monitoring and frequent arterial blood gas analysis thus ensuring a maximum of patient safety as well as precise and detailed records.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II to IV
* LVEF <= 45% (Echo within 28 days of enrollment)
* Predominantly central sleep apnea: AHI ≥15 events per hour, with >80% central events (apnoea or hypopnoea) and central AHI of ≥10 events per hour
* Peak VO2 < 90% of predicted value (CPX test within 28 days of enrollment) Nocturnal hypoxemic burden ≥ 25min/night
* Written informed consent

Exclusion criteria:

* Daytime hypercapnia (pCO2 > 45 mmHg)
* Ongoing ventilation therapy
* Severe COPD (chronic obstructive pulmonary disease) defined as FEV1< 50% (lung function test within 28 days of enrollment)
* Cardiothoracic surgery within the last 3 months
* Myocardial infarction within the last 6 months
* Unstable angina
* Acute myocarditis
* Stroke within the last 3 months
* Epilepsy or known cerebral damage or dementia
* Untreated restless-legs-syndrome
* Women of childbearing potential
* Participation in any clinical study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Reduction of hypoxemic burden | From date of enrolment until end of therapy phase (day 3). Hypoxemic burden is determined several times during this period.
  Reduction of hypoxemic burden >50% compared to baseline using oxygen-HFT versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bitter, MD, Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia
Locations (1):
- Heart and Diabetes Center North-Rhine-Westphalia, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No